CLINICAL TRIAL: NCT04833244
Title: Automatic Multimodal Assessment of Occurrence and Intensity of Pain for Research and Clinical Use
Acronym: MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manhattan Physical Medicine and Rehabilitation, LLP (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PRO00018713
Record Dates: First submitted 2017-05-07; First posted 2021-04-06 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Rotator Cuff Injuries
Keywords: Tree Number(s) C26.761.340 C26.803.063 C26.874.400; Unique ID D000070636
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled study in which the patient and investigator are blinded.
Who Masked: Participant, Outcomes Assessor
Masking Description: After qualifying, patients are randomized into intervention or control groups. The investigator and care provider then film the patient, teach the interventional or sham maneuver, and film the patient again. The outcomes assessor then evaluates the patient responses and filmed behaviors, but is not informed about whether the patient received the interventional maneuver or the sham maneuver.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Active Comparator): Patients are taught to draw their shoulders away from their heads and necks, activating the subscapularis and pectoralis muscles. When asked immediately afterwards to abduct and flex their shoulders, these muscles perform the action that generally engages the injured supraspinatus muscle, causing significant pain. However, when these muscles are substituted for the injured supraspinatus, abduction and flexion subsequently occur painlessly.
  Interventions: Behavioral: Triangular Forearm Support
- Control (Placebo Comparator): Patients are taught a sham maneuver that does little or nothing to alleviate the pain of abduction and flexion of the shoulders. Therefore their pain levels before and after learning the maneuver are likely to be similar.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Triangular Forearm Support — The intervention, the Triangular Forearm Support requires drawing the shoulders away from the subject's head and neck. This requires at least a mild force that this action can oppose. The most-favored maneuver is to have patients stand 2 feet away from a wall, interlock their fingers, and place their forearms to form two sides of an equilateral triangle against the wall. They then place their heads within the triangle, the backs of their heads close to or in on contact with the heels of their hands. Then, pressing against the wall with their elbows and forearms, they draw their shoulders as far away from the wall as possible, retaining contact between the wall and the tops of their heads. Subjects remain in this position for 45 seconds, at which time they stand erect and repeat the abduction and flexion maneuver.
  Other Names: Modified Dolphin Pose, Modified Headstand
  Arms: Interventional
Behavioral: Placebo — Patients will be asked to raise arms overhead for 45 seconds.
  Arms: Control

SUMMARY:
170 patients with rotator cuff syndrome will be filmed abducting and flexing their arms before learning a simple maneuver that alleviates most of the pain 90% of the time. They will then be filmed performing the same abduction and flexion of their arms. The patients will rate their pain on the common 10-point pain scale after abducting and flexing their arms before and after the maneuver.

DETAILED DESCRIPTION:
Facial expression and truncal metrics correlate strongly with occurrence and intensity of pain. Rotator cuff syndrome almost invariably gives significant pain, especially with abduction and flexion of the arms. A simple maneuver that alleviates that pain 90% of the time, by activating the subscapularis to perform the function of the damaged supraspinatus muscle. This study strives to correlate facial and truncal characteristics with the ten-point pain scale by correlating the filmed changes in facial and truncal characteristics with the variations in patient-rated pain before and after the pain-controlling maneuver.

Once effective, the maneuver may be repeated for a number of days, after which time patients generally remain pain-free permanently.

ELIGIBILITY:
Inclusion Criteria:

Rotator cuff syndrome -

Exclusion Criteria:

Psychological or emotional instability

Other orthopedic conditions of the shoulders

Cosmetic facial surgery

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between facial expression parameters and patient pain-scale ratings | Outcome measured within 1 minute of intervention
  Changes in facial muscular activity with changes in pain status
Reduction of pain in abduction and flexion following the triangular forearm support. maneuver. | Outcome measured within 1 minute of intervention
  Changes in Likert scale pain scores by patient and examinermaneuver abduction and flexion.

CONTACTS AND LOCATIONS:
Locations (1):
- Cara Cipriano, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] "Yoga-Based Maneuver Effectively Treats Rotator Cuff Syndrome." Fishman, Loren M.; Wilkins, Allen N.; Ovadia, Tova; Topics in Geriatric Rehabilitation . 27(2):151-161, April/June 2011.
- See also: Article describing efficacy of the TFS maneuver — http://journals.lww.com/topicsingeriatricrehabilitation/pages/results.aspx?txtkeywords=a+simple+maneuver